CLINICAL TRIAL: NCT07073911
Title: The Effect of a Group Exercise Intervention on Muscle Activation Patterns in People With Knee Osteoarthritis
Brief Title: Effect of Exercise on Muscle Activity, Strength, and Balance in People With Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gillian Hatfield (Other)
Collaborators: Les Mills International (Unknown)
Responsible Party: Sponsor-Investigator, Gillian Hatfield, Associate Professor, University of the Fraser Valley
Organization: University of the Fraser Valley (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101801
Record Dates: First submitted 2025-07-16; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Osteo Arthritis Knee and Hip
Keywords: muscle activity; gait; balance; strength
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise program (Experimental): Les Mills Thrive is a 45-minute class that consists of flexibility, strength, and coordination exercises designed to be delivered in a group fitness environment. Participants will have the option to attend group fitness classes in person, or do the exercise program at home on their own asynchronously, using recorded classes as guidance.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Les Mills Thrive is a 45-minute class that consists of flexibility, strength, and coordination exercises. This program aims to improve sensorimotor control and strength via functional weight-bearing exercises and floor exercises to isolate targeted hip and core muscles. In each class (whether in person or online), a certified Les Mills Thrive instructor will provide options to either increase or decrease the intensity of each exercise to cater to varying fitness levels and fluctuating symptoms. Each exercise has an assisted (using a chair for balance), body weight, and resisted (weight or exercise tubing) option. Participants will have the option to attend group fitness classes or do the classes asynchronously at home using a link to access a recorded class.
  Other Names: Les Mills Thrive

SUMMARY:
This will be a clinical trial of a standardized group exercise intervention, Les Mills Thrive, and determine if it alters muscle activation patterns and improves strength, balance, and symptoms in those with knee osteoarthritis (OA). Muscle activation patterns will be assessed using surface electromyography, strength will be assessed using isokinetic dynamometry, balance will be measured using the Community Balance and Mobility Scale (CB&M), and symptoms and typical activity will be measured using two questionnaires: the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), and the Physical Activity Scale for the Elderly (PASE). These outcome measures will be measured at baseline and after a 12-week group exercise intervention (Les Mills Thrive) for 42 older adults with knee OA. Results of this study will be disseminated via a report to Les Mills International, in community presentations, at relevant academic (e.g. Osteoarthritis Research Society International (OARSI) annual conference) and industry (e.g. Medical Fitness Association annual meeting) conferences, in an academic journal publication (e.g. Arthritis Care & Research), and through press releases or other media publications.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have received a diagnosis of knee OA from a physician and/or meet the American College of Rheumatology Clinical Classification Criteria for Osteoarthritis of the knee. The American College of Rheumatology criteria specify that a participant needs to have pain and fulfill three of the following six items: 1) aged 50 years or older, 2) no early morning stiffness or morning stiffness less than 30 minutes, 3) crepitus, 4) bony tenderness, 5) bony enlargement, 6) no palpable warmth
* They must pass the Get Active Questionnaire to ensure that they are safe to begin an exercise program (determined via recruitment email).

Exclusion Criteria:

* i) severe knee trauma, knee surgery, or intraarticular knee joint injections in the previous six months, ii) active synovitis, iii) concurrent neurological (i.e. Parkinson's disease, Alzheimer's dementia, or polyneuropathy), endocrine (i.e., diabetes mellitus) and/or vestibular disorders which may affect balance, iv) chronic disease that may put them at risk during the exercise classes (i.e., history of heart failure, stroke, chronic obstructive lung disease), v) uncorrected visual impairment which may affect balance, or vi) an inflammatory rheumatic disease (i.e., rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, and chronic reactive arthritis).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-08-26 (Estimated); Primary Completion 2026-06-19 (Estimated); Study Completion 2026-06-19 (Estimated)

PRIMARY OUTCOMES:
Quadriceps amplitude (Quadriceps PC1) | From initial data collection to the end of treatment at 12 weeks
  Surface electromyography (EMG) will be used to assess muscle activation patterns from the quadriceps and hamstrings. We will assess overall magnitude of activity as well as co-activation. These outcomes will be extracted from the EMG data using principal component analysis (PCA). PCA is a pattern recognition technique that extracts the main patterns in waveform data. It has previously identified patterns of quadriceps and hamstrings activity that are correlated with knee osteoarthritis progression. The first pattern extracted from quadriceps EMG waveforms (Quadriceps PC1) captures the overall magnitude (i.e. amplitude) of quadriceps activity.
Quadriceps co-activation ( Quadriceps PC2) | From baseline data collection to the end of the intervention at 12 weeks.
  Surface electromyography (EMG) will be used to assess muscle activation patterns from the quadriceps and hamstrings. We will assess overall magnitude of activity as well as co-activation. These outcomes will be extracted from the EMG data using principal component analysis (PCA). PCA is a pattern recognition technique that extracts the main patterns in waveform data. It has previously identified patterns of quadriceps and hamstrings activity that are correlated with knee osteoarthritis progression. The second pattern extracted from quadriceps EMG waveforms (Quadriceps PC2) captures prolonged quadriceps activity (i.e. co-activation).
Hamstrings amplitude (Hamstrings PC1) | From baseline data collection to the end of the intervention at 12 weeks.
  Surface electromyography (EMG) will be used to assess muscle activation patterns from the quadriceps and hamstrings. We will assess overall magnitude of activity as well as co-activation. These outcomes will be extracted from the EMG data using principal component analysis (PCA). PCA is a pattern recognition technique that extracts the main patterns in waveform data. It has previously identified patterns of quadriceps and hamstrings activity that are correlated with knee osteoarthritis progression. The first pattern extracted from hamstrings EMG waveforms (Hamstrings PC1) captures the overall magnitude (i.e. amplitude) of hamstrings activity.
Hamstrings co-activation (Hamstrings PC2) | From baseline data collection to the end of the intervention at 12 weeks.
  Surface electromyography (EMG) will be used to assess muscle activation patterns from the quadriceps and hamstrings. We will assess overall magnitude of activity as well as co-activation. These outcomes will be extracted from the EMG data using principal component analysis (PCA). PCA is a pattern recognition technique that extracts the main patterns in waveform data. It has previously identified patterns of quadriceps and hamstrings activity that are correlated with knee osteoarthritis progression. The second pattern extracted from hamstrings EMG waveforms (Hamstrings PC2) captures prolonged hamstrings activation (i.e. co-activation).

SECONDARY OUTCOMES:
Balance (Community Balance & Mobility Scale) | From baseline data collection to the end of the intervention at 12 weeks.
  The Community Balance and Mobility Scale (CB&M) was developed to assess community-level functional deficits in dynamic balance (locomotor stability during movement) and mobility. It assesses advanced balance and mobility activities such as rapid direction changes and dual tasking. This tool has been found to be valid and reliable in adults with knee OA , and avoids the ceiling effects of other balance tests like the Berg Balance Scale in individuals who can ambulate independently in the community.
Knee extensor strength | From baseline data collection until the end of the intervention at 12 weeks.
  Isometric knee extensor strength will be measured at 45 degrees of knee flexion using an isokinetic dynamometer. The participant will push as hard as they can against the dynamometer for 3 seconds. This will be repeated twice, with at least 2 minutes of rest between contractions.
Knee flexor strength | From baseline data collection until after the 12 week intervention.
  Isometric knee flexor strength will be measured at 55 degrees of knee flexion using an isokinetic dynamometer. The participant will push as hard as they can against the dynamometer for 3 seconds. This will be repeated twice, with at least 2 minutes of rest between contractions.
Symptoms (WOMAC) | From baseline data collection until after the 12 week intervention.
  Knee symptoms will be assessed using the Western Ontario & MacMaster Universities Osteoarthritis Index (WOMAC). This questionnaire assesses pain, stiffness, and function.
Physical activity | From baseline until after the 12 week intervention.
  Self-reported physical activity will be assessed using the Physical Activity Scale for the Elderly (PASE).

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Hatfield, PhD, Principal Investigator — University of the Fraser Valley
Locations (1):
- University of the Fraser Valley, Chilliwack, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Primary and secondary outcome measures: EMG data, balance scores, WOMAC scores, knee extensor and flexor strength, PASE scores
  Also participant age, sex, gender
Supporting Information: ICF
Time Frame: Approximately June 2026 until June 2031 (five years).
Access Criteria: Academics at other universities will be able to access the data by contacting the Primary Investigator via email.